CLINICAL TRIAL: NCT04908215
Title: A Randomised, Double-Blind, Vehicle-Controlled Phase 2 Study of Topically Applied INM-755 (Cannabinol) Cream in Patients With Epidermolysis Bullosa
Brief Title: INM-755 (Cannabinol) Cream for Treatment of Epidermolysis Bullosa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InMed Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 755-201-EB
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Epidermolysis Bullosa Simplex; Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa Dystrophica; Kindler Syndrome
MeSH Terms: conditions — Epidermolysis Bullosa Simplex; Epidermolysis Bullosa, Junctional; Epidermolysis Bullosa Dystrophica; Poikiloderma of Kindler | interventions — Cannabinol

STUDY DESIGN:
Intervention Model Description: Within-patient randomized, double-blind comparisons of INM-755 (cannabinol cream) versus vehicle cream (control) in matched, paired index areas
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: INM-755 (cannabinol cream) and vehicle cream (control) are identical in appearance and texture and packaged in kits labelled with unique blinded kit numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- INM-755 (cannabinol) cream (Experimental): Cannabinol cream, topically applied daily in thin layer on non-wound index areas and every 1, 2 or 3 days in thick layer on dressings for index wounds for a 28-day period.
  Interventions: Drug: INM-755 (cannabinol) cream
- Vehicle cream (Placebo Comparator): Vehicle cream, topically applied daily in thin layer on non-wound index areas and every 1, 2 or 3 days in thick layer on dressings for index wounds for a 28-day period.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: INM-755 (cannabinol) cream — topical cream containing cannabinol for dermal application
  Arms: INM-755 (cannabinol) cream
Drug: Vehicle Cream — topical cream base for dermal application containing no active agent
  Arms: Vehicle cream

SUMMARY:
The purpose of this study is to evaluate the safety of INM-755 (cannabinol) cream and obtain preliminary evidence of efficacy in treating symptoms and healing wounds over a 28-day period in patients with epidermolysis bullosa (EB).

DETAILED DESCRIPTION:
This is an international, multicenter study to evaluate the safety and obtain preliminary evidence of efficacy of topically applied INM-755 (cannabinol) cream in up to 20 patients with inherited EB (Simplex, Dystrophic, Junctional, or Kindler). The study uses a within-patient, double-blind design in which matched index areas are randomized to INM-755 (cannabinol) cream or vehicle cream as a control.

Selected index areas may be wounds or non-wound areas. Randomized treatments are applied daily to non-wound areas and every 1, 2, or 3 days on wounds, according to the patient's schedule for dressing changes. Treatment is over a 28-day period. EB symptoms are evaluated based on patient-reported outcomes. Wound healing is measured by digital photography. In this study designed to obtain preliminary evidence of efficacy, there is no single primary efficacy endpoint. Efficacy endpoints vary according to the presenting symptoms in each patient, which may include the presence of open wounds, wound pain associated with dressing changes, background wound pain (not procedurally linked), wound itch, and itch in non-wound areas. Net benefit from INM-755 cream is evaluated within each patient and based on their clinical needs at baseline.

Enrollment is beginning with adults and may be expanded to include adolescents.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female patients aged ≥18 years with documented diagnosis of any of the following types of inherited EB: Simplex, Junctional, Dystrophic, Kindler. Enrolment will be extended to patients ≥12 years old and <18 years old after positive opinion of a data monitoring committee after at least 4 adult patients have completed study.
* Presence of at least 1 pair of well-matched index areas. Up to 2 pairs of index areas (1 pair of non-wound and 1 pair of wound index areas) can be selected in each patient
* For non-wound itch index areas, both areas should:

  1. Have chronic itch with a score ≥40 mm on a 100 mm VAS
  2. Not exceed 20 percent of body surface area (BSA) or be less than 1 percent of BSA
  3. Be similar size, up to twice the area of the smaller index area
* For wound index areas, both wounds should:

  1. Have a surface area ≥5 cm^2 and ≤50 cm^2 inclusive and be aged ≥3 weeks
  2. Be well matched for size (up to twice the area of the smaller index area) and age (both either ≥3 weeks to 3 months or >3 months)
* Female patients of childbearing potential or men whose sexual partners are women of childbearing potential (WOCBP) must use highly effective birth control
* WOCBP must have a negative urine pregnancy test result at baseline
* Must provide written consent (or assent for patients aged <18 years with parental/guardian consent)

Key Exclusion Criteria:

* EB index areas have evidence of infection
* Patient has a systemic infection or used systemic antibiotics for EB-related infections within 7 days
* Use of systemic corticosteroids within 30 days or of topical corticosteroids on chosen index areas within 14 days
* Immunosuppressive therapy or cytotoxic chemotherapy within 60 days
* Use of any high potency opioid within 30 days
* Use of cannabis, cannabis extracts, or any cannabinoid products for medical or recreational use by any route of administration within 2 weeks
* Prior stem cell transplant or gene therapy for EB
* History of malignancy including basal cell and squamous cell carcinomas
* Arterial or venous disorder resulting in ulcerated wounds
* Uncontrolled diabetes mellitus
* Chronic pruritus primarily attributable to pathologies or conditions other than EB
* Blood transfusion to treat anemia within the past 3 months
* Use of any investigational drug within 30 days or 5 half-lives (whichever is longer)
* An underlying condition which places the patient at unacceptable risk
* Women who are pregnant, breastfeeding (lactating), or planning to become pregnant during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Non-Wound Itch by Visual Analogue Scale (VAS) | Baseline to Day 29
  Patients will report peak (maximal) pruritus intensity over the previous 24 hours using a 100 mm VAS (0 being "no itch" to 100 mm being "worst imaginable itch") recorded daily in the study diary. This outcome measure is applicable only for patients with non-wound index areas with eligible (moderate to severe) itch.
Change from Baseline in Wound Surface Area | Baseline to Day 29
  Wound surface area will be measured by digital photography at weekly intervals. This outcome measure is applicable only for patients with wound index areas.
Change from Baseline in Procedural Wound Pain by VAS | Baseline to Day 29
  Patients will report wound pain intensity using a 100 mm VAS (0 being "no pain" to 100 mm being "worst imaginable pain") and this will be recorded in the study diary. Procedural pain will be assessed immediately after each wound dressing, which may be every 1, 2, or 3 days according to an individual patient's schedule for dressing change. This outcome measure is applicable only for patients with wound index areas associated with eligible (moderate to severe) procedural pain.
Change from Baseline in Background Wound Pain by VAS | Baseline to Day 29
  Patients will report wound pain intensity using a 100 mm VAS (0 being "no pain" to 100 mm being "worst imaginable pain") and this will be recorded in the study diary. Peak (maximal) background pain will be assessed daily in the morning (done before the dressing change). This outcome measure is applicable only for patients with wound index areas associated with eligible (moderate to severe) background pain.
Change from Baseline in Wound Itch by VAS | Baseline to Day 29
  Patients will report peak (maximal) pruritus intensity over the previous 24 hours using a 100 mm VAS (0 being "no itch" to 100 mm being "worst imaginable itch") recorded daily in the study diary. This outcome measure is applicable only for patients with wound index areas associated with eligible (moderate to severe) itch.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra DJ Mancini, MSc, Study Director — InMed Pharmaceuticals Inc.
Locations (7):
- France (2):
  - Hopital Saint Louis APHP Paris, Paris
  - CHU Toulouse - Hopital Larrey, Toulouse
- Universitaetsklinikum Freiburg, Freiburg im Breisgau, Germany
- Andreas Syggros Hospital of Cutaneous Venereal Diseases, Athens, Greece
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Fondazione IRCCS Ca Granda. Ospedale Maggiore Policlinico, Milan, Milano
  - Instituto Dermopatico dell'Immacolata, IDI-IRCCS, Rome, Roma